CLINICAL TRIAL: NCT06570148
Title: Towards the Development of a Digital Solution to Support the Exchange of Information in Paediatric Rehabilitation: an Exploratory Qualitative Study With Professionals, Decision-makers and Patients Concerned : ProKidChildRehab
Brief Title: Stakeholder Perspectives on the Need for a Digital Solution in Pediatric Rehabilitation
Acronym: ProChRehab
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0029 - ProKChildRehab
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-03

CONDITIONS: Children; Disability Physical; Disabilities Multiple; Disability, Developmental
MeSH Terms: conditions — Developmental Disabilities | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-directed interview or focus group — Participants will be recruited using purposive sampling with maximum variation. If they meet the inclusion criteria, they will be invited to take part in an online interview or focus group, lasting between 40 minutes and 1.5 hours. During the Zoom interview or focus group, they will be asked to answer several pre-defined open-ended questions based on an interview grid co-constructed with the co-investigators, including a patient partner and parent partners. They will be asked to answer closed socio-demographic questions at the end of the interview or focus group. The Zoom meeting will be recorded (audio) and then transcribed into anonymized written form.

SUMMARY:
Introduction: Children with chronic conditions receive fragmented rehabilitative care due to the multitude of providers and structures involved, and the constant changes throughout their care and life course. E-health holds promise for supporting exchanges around the child and thus fostering more integrated care, but its adoption remains limited in healthcare settings.

Objective : the aim of this project is to explore the issues related to the usefulness and acceptability of a digital platform shared between children, their families and the professionals working with the children (rehabilitation, education, leisure) for monitoring children's health, to identify needs and preoccupations from the perspectives of the futur users, to inform the development of a digital application, named Deneo Kid.

Methodology: a qualitative study will be conducted. Semi-structured interviews will be conducted with professionals from the rehabilitation, education, social and leisure sectors in France, as well as decision-makers (healthcare executives, facility directors), and disabled children aged 11 to 25, to explore the opportunities, needs and concerns of these potential users with regard to this type of digital solution. The interviews will be conducted and recorded on Zoom. Only the audio recording will be kept, transcribed verbatim and then destroyed. At least 30 participants will be included, but it's when saturation is reached that the number of participants to be included will be determined. For the analysis, the 6 phases of a reflexive thematic analysis will be monitored using Nvivo12 software, by three analysts. The final themes will inform the development of a future digital health technology.

DETAILED DESCRIPTION:
In France, around 3 million children are carriers of a chronic disease. These children require individualized, highly specialized rehabilitation care supported by interdisciplinary teams, often over many years. Rehabilitation is defined as "a set of interventions designed to optimize the functioning and reduce the disability of people with health problems as they interact with their environment". The main objective of rehabilitation is thus to promote the child's social participation in his or her daily life, whether at home, school or leisure. To achieve this goal, the partnership between all the professionals involved with the child, the child and his or her family is essential. The exchange of information between these stakeholders must be optimal throughout the child's care. However, there are many gaps in access to and sharing of information around the child, due to the multiplicity of stakeholders involved, the constant changes (care structures, school, etc.) and the wide variety of contexts (school, home, private practice, leisure, hospital). E-health or digital health presents multiple opportunities to promote access to information, improve monitoring of children, involve the family in care and reduce the mental burden associated with information exchanges, which are mainly handled by the family. The Deneo KID project, led by W.Inn, Brest University Hospital's innovation center, and carried out in partnership with the Deneo company, aims to meet these challenges. It aims to develop a digital solution for exchanging information between the various players involved in the child's care. This study is therefore directly in line with the Deneo KID project.

Indeed, it is recognized in the literature that taking into account the needs and expectations of users (families, professionals, children) from the earliest design phases of a digital solution is essential to foster its usability, acceptability and future appropriation by its users. But this is not enough, and the literature shows a high percentage of failure in digital health innovation projects. For a solution to be adopted by its users, it is also essential to take into account the obstacles and brakes to the implementation of this type of solution at different levels (professionals, decision-makers). Indeed, authors have highlighted organizational factors likely to hinder or support the adoption of this type of solution, such as organizational support, or the persuasive strategies and techniques implemented by the organization to encourage the adoption of a solution by the professionals on a team.

Considering these elements, the investigators have chosen to include not only people concerned by the use of the solution, but also people empowered to lead change, i.e. decision-makers in settings welcoming children with chronic health conditions. Decision-makers is defined as those involved in decision-making concerning the implementation of digital solutions in the various structures working for the health of children with chronic health conditions. They may be health managers or senior health managers in hospitals and rehabilitation centers, directors or heads of department in medico-social establishments, or association leaders. This will enable us to work with decision-makers to define appropriate implementation strategies to encourage adoption of the solution in care environments, and thus guarantee the success of the Deneo KID project.

A qualitative focus group study of families of children with chronic illnesses was already carried out in 2022, supported by the Ildys Foundation (PITChREHAB study). Its aim was to explore the needs and expectations of families of children with chronic illnesses with regard to digital solutions to promote the exchange of information related to their child's rehabilitation. This study highlighted multiple opportunities for families, as well as essential functionalities to be included in the future Deneo KID solution from the families' point of view.

The ProChildRehab study is the second stage in the development of the Deneo KID solution. It focuses on the needs of child-facing professionals and decision-makers for a digital solution designed to facilitate the exchange of information about children with disabilities.

The ProChildRehab study is the second stage in the development of the Deneo KID solution. It focuses on the needs of professionals working with children and decision-makers for a digital solution designed to facilitate the exchange of information about children with disabilities.

The ProChildRehab study was approved by the CHU de Brest territory ethics committee on 14/03/2024. Since then, interviews have been carried out with 18 health, education and leisure professionals working with children with disabilities (psychologist, PRM doctor, specialist teacher, AESH, Handisport leader, etc.) and 6 decision-makers (health executive, SESSAD director, Handisport manager, etc.). Further interviews are planned, as data saturation has not yet been reached (there is some redundancy in the answers, but new ideas are still being contributed). Analysis of these interviews is underway (an iterative process in qualitative research, with analysis concurrent with data collection). Initial results suggest that the views of patients concerned by this future digital solution should be taken into account. Indeed, there is no consensus on several points, such as the psychological information that could be shared by the child and his parents with professionals via the platform (e.g. the child's morale), the fact of sharing photos of daily life and therefore quite intimate (e.g. photos of the house), the usefulness of proposing self-rehabilitation exercises to patients via the platform (rehabilitation overload for children vs. ensuring continuity of services), or the perception of what the child's "reality" is (e.g. professionals who ask for more information on the child's reality to better support him/her vs. other professionals who say that this information is confidential). The investigators would therefore like to explore with young people the acceptability of certain features, particularly in terms of the information that is acceptable for them to exchange about their health via this platform. The aim is to question people who could be concerned by the sharing of information through this future solution, i.e. young people with disabilities who are living or have lived through the care of a child with a disability.

These initial data obtained and the need to go out and interview patients corroborate with the literature on the subject, which highlights the gaps between patients' and clinicians' perceptions of their needs and interests with regard to e-health and advocates an "alignment of concerns" on both sides.

ELIGIBILITY:
PROFESSIONALS

Inclusion Criteria :

* Be a health, social, educational or leisure professional involved in the rehabilitation of children with disabilities (doctor, physiotherapist, occupational therapist, kinesiologist, psychomotor therapist, speech therapist, psychologist, specialized educator, social worker, school nurse, sports educator in a leisure center, nursery assistant in a crèche, etc.).
* Speak and understand French

DECISION MAKERS

Inclusion Criteria:

* Be a professional working in the health or social field and managing or coordinating a team of rehabilitation professionals working in pediatrics (clinical coordinator, health executive, senior health executive, clinical expert, director of a medico-social establishment, etc.), or a leisure structure for children with disabilities, or a crèche for children with disabilities.
* Speak and understand French

PATIENTS

Inclusion criteria:

* be between the ages of 11 and 25
* have had a disability as defined by the International Classification of Functioning and Disability (ICF) since childhood
* have undergone or be undergoing paediatric rehabilitation care
* have been followed or be followed by at least 3 different rehabilitation, school or leisure professionals (e.g. private physiotherapist, APA Handisport, specialized school teacher, etc.)
* have good oral communication skills

Exclusion criteria:

- communication difficulties (e.g. aphasia) or intellectual deficiencies that make it impossible to express oneself during an interview lasting about 1 hour

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Professionals: a health, social, educational or leisure professional involved in the rehabilitation of children with disabilities (doctor, physiotherapist, occupational therapist, kinesiologist, psychomotor therapist, speech therapist, psychologist, specialized educator, social worker, school nurse, sports educator in a leisure center,...)
  Decision-makers: a professional working in the health or social field and managing or coordinating a team of rehabilitation professionals working in pediatrics (clinical coordinator, health executive, senior health executive, clinical expert, director of a medico-social establishment, etc.), or a leisure structure for children with disabilities,...)
  Patients: young people aged 11 to 25 living with a disability
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
List of needs for the future app : list of needs expressed by professionals, decision-makers and patients with regard to priority information exchanges via digital solutions | 24 months
  This outcome will be collected qualitatively, using open-ended questions asked during a semi-structured individual interview with each participant. Their needs will be explored using open-ended and follow-up questions (e.g.: what are your needs for information exchange with the family? with the child? with other professionals? how could a digital solution facilitate these exchanges?)
  A qualitative analysis (inductive) will help to meet this outcome
List of facilitators and barriers of the app adoption : List of facilitators and barriers of digital health technology adoption among health professionals, decision makers and patients | 24 months
  This outcome will be collected qualitatively, using open-ended questions asked during a semi-structured individual interview with each participant. Their needs will be explored using open-ended and follow-up questions (e.g.: what concerns do you have about using a digital solution to communicate with the family? with the child? with other professionals? what do you think would facilitate adoption of the solution in your environment?)
  A hybrid qualitative analysis (inductive and deductive using an implementation science model such as the CFIR, Damschroder et al., 2022 will help to meet this outcome)
List of strategies to implement the app : List of strategies to implement digital health technology in a pediatric rehabilitation context, from the perspectives of different end users | 24 months
  This outcome will be collected qualitatively, using open-ended questions asked during a semi-structured individual interview with each participant. Their needs will be explored using open-ended questions and follow-up questions (e.g.: what would be the key determinants for such a solution to be implemented in your area? What strategies at micro/meso/macro level?)
  A hybrid qualitative analysis (inductive and deductive using an implementation science model such as the CFIR, Damschroder et al., 2022 will help to meet this outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Kersalé, Principal Investigator — CHU de Brest
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Kersale M, Hong QN, Richard T, Kandalaft Cabrol C, Guevel A, Fily E, Tisserand G, Brochard S, Pomey MP, Pons C. Perspectives From Multidisciplinary Professionals in France on Shared Patient Portals for Integrated Pediatric Rehabilitation: Qualitative Study. JMIR Rehabil Assist Technol. 2025 Oct 10;12:e73068. doi: 10.2196/73068. PMID 41072921